CLINICAL TRIAL: NCT03445468
Title: Phase III Study to Evaluate Immunogenicity and Safety of 'Il-Yang Quadrivalent Seasonal Influenza Vaccine' in Healthy Korean Children and Adolescents
Brief Title: Immunogenicity and Safety for 'IL-YANG Quadrivalent Influenza Vaccine' in Healthy Korean Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IF4CH03
Record Dates: First submitted 2017-08-08; First posted 2018-02-26 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2018-08

CONDITIONS: Influenza, Human
Keywords: Influenza vaccine; Split influenza vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-YANG Quadrivalent Influenza Vaccine (Experimental): The vaccine contains both B strain (Yamagata, Victoria)
  Interventions: Biological: IL-YANG Quadrivalent Influenza Vaccine
- IL-YANG Flu Vaccine Pre-filled Syringe (Active Comparator): The vaccine contains the B/Yamagata strain and it was approved for commercial sale by Ministry of Food and Drug Safety.
  Interventions: Biological: IL-YANG Flu Vaccine Pre-filled Syringe

INTERVENTIONS:
Biological: IL-YANG Quadrivalent Influenza Vaccine — A single 0.5mL dose administrated as an intramuscular injection.
  Arms: IL-YANG Quadrivalent Influenza Vaccine
Biological: IL-YANG Flu Vaccine Pre-filled Syringe — A single 0.5mL dose administrated as an intramuscular injection.
  Arms: IL-YANG Flu Vaccine Pre-filled Syringe

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of 'IL-YANG Quadrivalent Seasonal Influenza Vaccine' in healthy Korean children and adolescents.

DETAILED DESCRIPTION:
The study is an open-label(Part 1), Single-arm(Part 1), Randomized(Part 2), Double-blind(Part 2), Active comparator(Part 2) Phase III study.

Before initiation of any protocol-specific activities, written informed consent is obtained from each patient and their legally acceptable representatives. Subjects who meet all of the eligibility criteria after screening assessments as specified in the protocol, are randomized into the test group or the comparator group in a ratio of 4 :1 and receive a single dose or two doses of the study vaccine. The investigator perform the efficacy (immunogenicity) and safety assessments throughout the study. Efficacy data are collected at Visit 1 (prior to vaccination) and at the end-of-study visit for efficacy (immunogenicity) assessments, and for safety assessment, subjects and their legally acceptable representatives are instructed to record any treatment-emergent adverse event in Patient Diary cards.

For all randomized subjects, blood sample is obtained prior to vaccination, and the study vaccine 0.5mL is administered. For children aged from 3 years to <9 years of age who have not previously received influenza vaccine, another dose of the study vaccine is administered 4 to 5 weeks after the first dose. Blood samples are collected 4 to 5 weeks after the last dose of the study drug for the assessment of antibody titer. All subjects are followed for 6 months after the last dose of the study drug for the safety assessments, and Month 6 follow-up visit is the end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged from 3 years to < 19 years
* Subjects were born after full term pregnancy (37 weeks)
* Woman of childbearing potential must have a negative result from Urine Human Chorionic Gonadotropin(HCG) test at the screening visit.
* Voluntary written informed consent was obtained from the subject and the subject's legally acceptable representative (consent of legally acceptable representative was required for subjects younger than 7 years of age)

Exclusion Criteria:

* Subject with a known serious allergy reaction after influenza vaccination or to any component vaccine including eggs
* Subject who had received an influenza vaccine within the last 6 months
* Subject who has, or has a family history of, an immune system disorder including immune deficiency disease
* Subject with a history of Guillain-Barre syndrome
* Subject with Down's syndrome or cytogenetic disorders.
* Subject with severe chronic disease which in the investigator's opinion would not make the subject a good candidate for the clinical trial
* Subject with hemophilia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subject who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine
* Subject who had previously received another vaccine within 28 days before administration of the study drug, or is scheduled to receive another vaccine during the study period.
* Subject who had received immunosuppressant or immune modifying drug within the last 3 months prior to administration of the study vaccine
* Subject who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or is expecting to be treated with immunoglobulin or blood-derived products during the study.
* Subject who had participated in another experimental study within 28 days prior to administration of the study vaccine
* Subject with other clinically significant medical or psychological condition who in the investigator's opinion would not be suitable for the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 379 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate against Hemagglutination Inhibition(HI) antibody | Up to Day28(+7) after the last vaccination
  Seroconversion rate(a lower bound of 95 CI) ≥ 40%
Seroprotection rate against Hemagglutination | Up to Day28(+7) after the last vaccination
  Seroprotection rate(a lower bound of 95 CI) ≥ 70%

SECONDARY OUTCOMES:
Geometric Mean Titer(GMT) and Geometric Mean Ratio(GMR) | Up to Day28(+7) after the last vaccination
  GMT and GMR of HI Antibody Titer Before Vaccination and After Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Han Kang, MD.PhD, Principal Investigator — The catholic university of Korea, Seoul ST. Marry's Hospital
Locations (1):
- The catholic university of Korea, Seoul ST. Marry's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No